CLINICAL TRIAL: NCT06215755
Title: A Phase 1b, Open-Label, Multiple Ascending Dose, Multicenter Study of VRG50635 in Participants With Sporadic and Familial Amyotrophic Lateral Sclerosis Followed by Long-Term Treatment
Brief Title: A Study of VRG50635 in Participants With Amyotrophic Lateral Sclerosis (ALS)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Study terminated by Sponsor due to lack of risk-benefit data.
Sponsor: Verge Genomics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VGCS-50635-002; 2023-506509-21 (EudraCT Number)
Record Dates: First submitted 2023-12-18; First posted 2024-01-22 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: VRG50635; Familial Amyotrophic Lateral Sclerosis; Sporadic Amyotrophic Lateral Sclerosis; ALS
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Amyotrophic lateral sclerosis 1

STUDY DESIGN:
Intervention Model Description: Part 1, no study drug will be administered.
  Part 2, the starting dose is 400 mg for 8 weeks (Treatment Period 1) and doses will be escalated to 600 mg for 8 weeks (Treatment Period 2) and 800 mg for 8 weeks (Treatment Period 3).
  Part 3, each participant will continue receiving treatment with the highest tolerated dose achieved in Part 2 for up to 40 weeks.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VRG50635 (Experimental): The study drug is VRG50635 200 mg oral capsules. VRG50635 will be administered as oral capsules once daily in the morning after a low-fat meal, approximately 30 minutes prior to VRG50635 administration. Following administration there is a 5 to 6-hour restriction period where participants should consume only low-fat food.
  Interventions: Drug: VRG50635

INTERVENTIONS:
Drug: VRG50635 — Part 1, no study drug will be administered.
  Part 2, the starting dose is 400 mg for 8 weeks (Treatment Period 1) and doses will be escalated to 600 mg for 8 weeks (Treatment Period 2) and 800 mg for 8 weeks (Treatment Period 3).
  Part 3, each participant will continue receiving treatment with the highest tolerated dose achieved in Part 2 for up to 40 weeks.

SUMMARY:
The primary purpose of this study is to evaluate the safety and tolerability of VRG50635 in participants with ALS.

DETAILED DESCRIPTION:
This is a Phase 1b, open-label, within-participant, multiple ascending dose, multicenter study of VRG50635 in participants with sporadic amyotrophic lateral sclerosis (sALS) and familial amyotrophic lateral sclerosis (fALS). Part 1 is a pre-treatment run-in period to establish the mean baseline based on repeated measurements of all biomarkers in eligible participants prior to initiating dosing with VRG50635. In Part 2, the safety, tolerability, PK, and efficacy of VRG50635 will be evaluated using a within-participant multiple ascending dose scheme. In Part 3, the long-term tolerability, safety, and efficacy of VRG50635 will be evaluated at the highest tolerated dose.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent and be willing and able to comply with the requirements of the study protocol.
2. Must be ≥ 18 and ≤ 75 years of age at the time of signing the informed consent form (ICF).
3. Have a diagnosis of ALS according to the Gold Coast Diagnostic Criteria.
4. Have either sporadic amyotrophic lateral sclerosis (sALS) or familial amyotrophic lateral sclerosis (fALS).
5. Treatment Research Initiative to Cure ALS (TRICALS) risk profile > -6.00 and < -2.00.
6. Have slow vital capacity (SVC) ≥ 60% of the predicted value.
7. Have a score of 3 or 4 on Item #3 (Swallowing) of the Harmonized ALS Functional Rating Scale-Revised (ALS-FRS-R). Participants with a score of 3 can be enrolled with the Sponsor's approval only if they are able to safely swallow capsules.
8. Have a body weight ≥ 45 kg and body mass index (BMI) ≥ 18 kg/m2.
9. Participants of childbearing potential are eligible to participate if they are not pregnant or breastfeeding and agree to use one highly effective method of contraception, if sexually active, for the duration of the study through 90 days after the last study drug administration. Participants must not donate eggs for the duration of study through 90 days after the last dose of study drug.
10. Participants capable of producing sperm and their partners of childbearing potential must agree to use condoms and one highly effective method of contraception, respectively, for the duration of the study through 90 days after the last study drug administration. Participants must not donate sperm for the duration of study through 90 days after the last dose of study drug.
11. Be able and willing to undergo measurement of at-home mobility using contactless sensors connected to the internet.
12. Be able and willing to have clinic or at-home visits during the study.

Exclusion Criteria:

1. Have active psychiatric disease, substance abuse, neuromuscular weakness other than ALS, or any other medical condition that, in the opinion of the Investigator, might confound the results of the study or interfere with the intake or absorption of the study drug or participation for the full duration of the study.
2. Have a history of unstable or severe cardiac, pulmonary, neurological, oncological, hepatic, or renal disease or another medically significant illness other than ALS precluding their safe participation in this study.
3. Have a history of substance use disorder or illicit drug use in the last year (medically prescribed or over-the-counter cannabis use is allowed, if legal in the country).
4. Have a history of serious infection (e.g., pneumonia, septicemia) ≤ 4 weeks of Screening; infection requiring hospitalization or treatment with intravenous (IV) antibiotics, antivirals, or antifungals within 4 weeks of Screening; or chronic bacterial infection (e.g., tuberculosis) deemed unacceptable as per the Investigator's judgment.
5. Had major surgery ≤ 4 weeks before Screening.
6. Be currently taking or planning to take strong cytochrome P450 3A4 (CYP3A4) inhibitors or inducers.
7. Be currently taking or have discontinued treatment with riluzole < 4 weeks before Screening. Participants who have been taking a stable dose of riluzole for ≥ 4 weeks are eligible if they remain on the same dose throughout the duration of the study.
8. Be taking Radicava (administered orally or IV as approved in the participant's country), Relyvrio, any other approved standard of care treatment, or tauroursodeoxycholic acid (TUDCA) as a dietary supplement administered for < 4 weeks prior to Screening or on a schedule of treatment different from the approved standard schedule of treatment. Participants who have completed ≥ 4 weeks of treatment before Screening are eligible if they plan to continue treatment at a stable dose throughout the duration of the study.
9. Have an active malignancy or history (≤ 1 years prior to enrollment) of solid, metastatic, or hematologic malignancy. Exception: basal cell carcinoma in situ of the skin that has been adequately treated.
10. Be diagnosed with long QT syndrome. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointes) should be discussed with and approved by the study medical monitor prior to enrollment.
11. Have a prolonged corrected QT interval using Fridericia's formula (QTcF) at the Screening visit ECG > 450 ms for male participants and > 470 ms for female participants.
12. Have an active SARS-CoV-2 infection or positive COVID-19 test at Screening.1
13. Have one or more of the following laboratory test abnormalities at Screening: (a) Positive hepatitis C virus (HCV) antibodies with confirmation by HCV-RNA polymerase chain reaction (PCR) reflex testing; (b) Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). Note: If a participant is negative for HBsAg but positive for HBcAb, the participant is eligible if the participant tests positive for the antibody to HBsAg reflex testing.
14. Have uncontrolled seizures.
15. Have a documented history of attempted suicide within 6 months prior to the Screening visit, or suicidal ideation of category 4 or 5 on the screening Columbia-Suicide Severity Rating Scale (C-SSRS), or be at significant risk for suicide, in the opinion of the Investigator.
16. For participants of childbearing potential, be pregnant or breastfeeding.
17. Have received a live vaccine within 14 days before Screening.
18. Be concurrently participating in any other interventional clinical study or have received treatment with another investigational drug within 4 weeks or 5 half-lives of the investigational agent before the Screening visit, whichever is longer. Participation in observational studies is allowed.
19. Have received stem cell or gene therapy for ALS at any time in the past.
20. At the Screening visit, have one or more of the following:

    1. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 3.0 × upper limit of normal (ULN)
    2. Bilirubin > 1.5 × ULN, unless the participant has documented Gilbert syndrome (isolated bilirubin > 1.5 × ULN is acceptable if bilirubin is fractionated and direct bilirubin is < 35%)
    3. Serum albumin < 3 g/dL
    4. Hemoglobin < 9.0 g/dL
    5. Platelets < 30,000/μL
    6. Estimated glomerular filtration rate < 90 mL/min/1.73 m2 (Modification of Diet in Renal Disease [MDRD])

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2024-01-15 (Actual); Primary Completion 2025-07-07 (Actual); Study Completion 2025-07-07 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment-emergent Adverse Events (TEAEs) | Up to 80 weeks
Number of Participants with Clinical Laboratory Evaluation Abnormalities | Up to 80 weeks
Number of Participants with Vital Sign Abnormalities | Up to 80 weeks
Number of Participants with Electrocardiogram (ECG) Abnormalities | Up to 80 weeks
Number of Participants with Physical Examination Abnormalities | Up to 80 weeks
Number of Participants with Neurological Examination Abnormalities | Up to 80 weeks

SECONDARY OUTCOMES:
Maximum Observed Concentration (Cmax) | Up to 80 weeks
Area Under the Concentration-time Curve (AUC) | Up to 80 weeks
Time to Maximum Observed Concentration (tmax) | Up to 80 weeks
Change from Baseline in Plasma Levels of Neurofilament Light Chain (NfL) as Measured by Immunoassay | Baseline, up to 80 weeks
Time to Disease Progression | Up to 80 weeks
Change in Harmonized ALS Functional Rating Scale-Revised (ALS-FRS-R) Score | Up to 80 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Diego Cadavid, MD, Study Director — Verge Genomics
Locations (7):
- UZ Leuven, Leuven, Flemish Brabant, Belgium
- Canada (2):
  - Stan Cassidy Centre for Rehabilitation (Horizon NB), Montreal, Quebec
  - The Neuro - Montréal Neurological Institute-Hospital, Montreal, Quebec
- Finland (3):
  - University of Eastern Finland, Brain Research Unit, Kuopio, Eastern Finland
  - Helsinki University Hospital, Helsinki, Uusimaa
  - Turku University Hospital, Turku, Western Finland
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hung ST, Linares GR, Chang WH, Eoh Y, Krishnan G, Mendonca S, Hong S, Shi Y, Santana M, Kueth C, Macklin-Isquierdo S, Perry S, Duhaime S, Maios C, Chang J, Perez J, Couto A, Lai J, Li Y, Alworth SV, Hendricks E, Wang Y, Zlokovic BV, Dickman DK, Parker JA, Zarnescu DC, Gao FB, Ichida JK. PIKFYVE inhibition mitigates disease in models of diverse forms of ALS. Cell. 2023 Feb 16;186(4):786-802.e28. doi: 10.1016/j.cell.2023.01.005. Epub 2023 Feb 7. PMID 36754049
- [Background] Shi Y, Lin S, Staats KA, Li Y, Chang WH, Hung ST, Hendricks E, Linares GR, Wang Y, Son EY, Wen X, Kisler K, Wilkinson B, Menendez L, Sugawara T, Woolwine P, Huang M, Cowan MJ, Ge B, Koutsodendris N, Sandor KP, Komberg J, Vangoor VR, Senthilkumar K, Hennes V, Seah C, Nelson AR, Cheng TY, Lee SJ, August PR, Chen JA, Wisniewski N, Hanson-Smith V, Belgard TG, Zhang A, Coba M, Grunseich C, Ward ME, van den Berg LH, Pasterkamp RJ, Trotti D, Zlokovic BV, Ichida JK. Haploinsufficiency leads to neurodegeneration in C9ORF72 ALS/FTD human induced motor neurons. Nat Med. 2018 Mar;24(3):313-325. doi: 10.1038/nm.4490. Epub 2018 Feb 5. PMID 29400714